CLINICAL TRIAL: NCT04304222
Title: Application of 3D Printed Removable Denture Prosthesis Framework for Partial Edentulous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Dental Centre, Singapore (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SHF/FG701S/2017
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Dental Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Participants are randomized into 2 sequence:
  1. To receive the conventionally made denture framework then the 3D printed denture framework
  2. To receive the 3D printed denture framework then the conventionally made denture framework
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 2 study team clinicians are the designated care providers to the participants hence they are masked together with the participants. One of the masked clinicians is the Principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Other): To receive the conventionally made denture framework then the 3D printed denture framework.
  Interventions: Device: 3D Printed Denture Framework
- Sequence B (Other): To receive the 3D printed denture framework then the conventionally made denture framework.
  Interventions: Device: 3D Printed Denture Framework

INTERVENTIONS:
Device: 3D Printed Denture Framework — The Denture Framework is 3D printed from the digital image obtained from the denture mold.

SUMMARY:
Tooth loss is a major dental problem worldwide. A recent study in Singapore found that approximately one third of adults aged over 65 are living without any natural teeth. Prevalence of loss of some teeth, or partial edentulism, in this population is estimated to be even higher. Tooth loss has a series of deleterious consequences for oral and general health. The high prevalence of tooth loss has resulted in great needs and demands of prosthetic replacements, posing challenges to the public dental care system in Singapore. Removable dentures are the most widely and commonly used device to replace missing teeth and restore oral functions. The removable denture possesses a metal framework that connects other components of the denture, to ensure rigidity and stability while in function. However, the current method of fabricating denture frameworks is a complex, error-prone, time-consuming, and expensive process. Due to the inherent inaccuracies in the materials and technique, fit of the framework is compromised and undesirable to meet patients' satisfaction. With the new development of computer aided design and 3D printing metal techniques, it is now possible to apply digital design and manufacturing for the fabrication of dentures. This proposal aims to compare the precision and fit, and patient satisfaction, of 3D printed and conventional casted removable denture frameworks in preclinical and clinical settings.

DETAILED DESCRIPTION:
Tooth loss or edentulism is a major dental problem worldwide, particularly among the senior population. A recent study in Singapore found that approximately one third of adults aged over 60 are living with complete edentulism. Prevalence of partial edentulism in this population is estimated to be even higher. The high prevalence of tooth loss has resulted in great needs and demands of prosthetic replacements, posing challenges to the public dental care system in Singapore. Removable denture prosthesis is the most commonly used device to replace missing teeth and restore oral functions. The removable denture prosthesis possesses a metal framework that connects the clasps, retainers, base and acrylic teeth, to ensure rigidity and stability while in function. However, the current way of fabricating denture frameworks using casting method is a time consuming, complex, error-prone, and expensive process. Due to the inherent inaccuracies in the materials and technique, the fit of the framework is compromised and undesirable to meet patients' satisfaction. With recent developments in computer aided design and additive manufacturing, commonly known as 3D printing or rapid prototyping, the techniques allow for printing of complex metal structures of high strength, stiffness and chemical resistance. This proposal aims to compare the precision and fit, and patient's satisfaction, of 3D printed denture frameworks and eventually translate this to a more efficient denture fabricating process.

The removable denture prosthesis is the most commonly used device to replace missing teeth and restore oral functions in patients with partial and complete edentulism. The fabrication of framework using conventional methods is time consuming and inaccurate. Thus the ultimate goal of this study is to enhance the workflow efficiency, improve the fabrication precision of the device, reduce treatment cost and time, and promote oral function and overall quality of life of patients. At the same time, the research methods developed from this study is a platform for the study of new dental devices, with potential applications for new digital dental practices. Thus, if successful, the deliverables from this research will both advance dental research, and extend applicable knowledge to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partial edentulism requiring RDPs
* Above the age of 21 years
* Medically fit
* Prior denture experience

Exclusion Criteria:

* New denture wearers
* Patients with a history of maladaptation to denture use
* Patients with maxillofacial defects

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
To compare the space between the occlusal rest and the corresponding rest seat among the 3D printed and conventional fabricated removable dental prosthesis (RDP) frameworks in partial edentulous patients. | End of study
  The space between the occlusal rest and the corresponding rest seat in 3D printed framework is smaller than the casting framework.

SECONDARY OUTCOMES:
To compare the patients' satisfaction towards the use of 3D printed and conventional casting RDP frameworks. | End of study
To compare the space between the occlusal rests, clasps and minor connectors of 3D printed and conventional casting RDP frameworks on patient models in the dental lab. | End of study

CONTACTS AND LOCATIONS:
Locations (1):
- National Dental Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No